CLINICAL TRIAL: NCT04740723
Title: A Renal Artery Denervation Feasibility Study of the MetAvention Integrated Radio Frequency Denervation System for the Treatment of Hypertension
Brief Title: Evaluation of the Integrated Radio Frequency Denervation System for the Treatment of Hypertension
Acronym: RADAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metavention (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 1880
Record Dates: First submitted 2021-01-25; First posted 2021-02-05 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Hypertension; Metabolic Syndrome
Keywords: Renal Denervation
MeSH Terms: conditions — Hypertension; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: The study is a prospective, single-arm, multi-center, non-randomized feasibility trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Renal denervation (Experimental): Renal denervation with the iRF system
  Interventions: Device: iRF System Renal Denervation

INTERVENTIONS:
Device: iRF System Renal Denervation — The iRF System is a percutaneous, catheter-based device which uses RF energy to circumferentially denervate the sympathetic nerves surrounding the artery

SUMMARY:
The objective of the study is to evaluate the safety of renal denervation using the iRF System and to understand any potential improvement in hypertension.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, multi-center, non-randomized trial to evaluate the initial safety and performance of renal denervation with the iRF system for the treatment of hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 80 years old
2. Office SBP ≥ 140 and < 180 mmHg on a stable dose of antihypertensive medication(s) for at least 30 days
3. Documented daytime systolic ABP ≥ 135 and < 170 mmHg
4. Waist circumference ≥ 102 cm (male) and ≥ 88 cm (female)

   Exclusion Criteria:
5. Renal artery anatomy on either side, ineligible for treatment including the following:

   1. Main renal artery diameter < 4.0 mm or > 7.0 mm
   2. Main renal artery length < 20.0 mm
   3. Only one functioning kidney
   4. Presence of abnormal kidney tumors
   5. Renal artery with aneurysm
   6. Pre-existing renal stent or history of renal artery angioplasty
   7. Fibromuscular disease of the renal arteries
   8. Presence of renal artery stenosis of any origin ≥ 30 %
   9. Individual lacks appropriate renal artery anatomy
6. Prior renal denervation procedure
7. Iliac/femoral artery stenosis precluding insertion of the iRF Catheter
8. Evidence of active infection within 7 days of the Index Procedure
9. Type 1 diabetes mellitus
10. Documented history of chronic active inflammatory bowel disorders such as Crohn disease or ulcerative colitis
11. eGFR < 45 mL/min per 1.73 m2
12. Brachial circumference ≥ 42 cm
13. Any history of cerebrovascular event (e.g., stroke, transient ischemic event, and cerebrovascular accident) within 6 months of patient consent
14. Myocardial infarction within 6 months of patient consent
15. Heart failure (New York Heart Association [NYHA] Class III-IV) at time of consent
16. Documented confirmed episode(s) of stable or unstable angina within 6 months of patient consent
17. Documented history of persistent or permanent atrial tachyarrhythmia
18. Chronic oxygen support or mechanical ventilation other than nocturnal respiratory support for sleep apnea
19. Night shift workers
20. Chronic regular use (e.g., daily use) of NSAIDs for 6 months or greater. Aspirin therapy is allowed.
21. Active implantable medical device (e.g., ICD or CRT-D, neuromodulator/spinal stimulator, baroreflex stimulator)
22. Primary pulmonary HTN (> 60 mmHg pulmonary artery or right ventricular systolic pressure)
23. Individual has known pheochromocytoma, Cushing syndrome, primary hyperaldosteronism, coarctation of the aorta, untreated hyperthyroidism, untreated hypothyroidism, or primary hyperparathyroidism. (Note: Treated hyperthyroidism and treated hypothyroidism are permissible.)
24. Documented contraindication or allergy to contrast medium not amenable to treatment
25. Limited life expectancy of < 1 year at the discretion of the investigator
26. Any known, unresolved history of drug use or alcohol dependency, lacks the ability to comprehend or follow instructions, or for any reason in the opinion of the investigator, would be unlikely or unable to comply with study protocol requirements or whose participation may result in data analysis confounders (e.g., night shift workers)
27. Pregnant, nursing, or planning to become pregnant (documented negative pregnancy test result required documented within a maximum of 7 days before procedure for all women of childbearing potential)
28. Concurrent enrollment in any other investigational drug or device trial (participation in noninterventional registries is acceptable)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-06 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
Rate of Major Adverse Events | Index Procedure through 30 days
  Incidence of the following Major Adverse Events (MAEs)
  * Death (all-cause)
  * New onset end stage renal disease
  * Significant embolic events resulting in end-organ damage
  * Renal artery perforation or dissection requiring intervention
  * Hospital admission for hypertensive crisis not related to confirmed non-adherence with medications or protocol
  * New renal stenosis > 70 %

SECONDARY OUTCOMES:
Change in Systolic/Diastolic Blood Pressure - Average Automated Office Blood Pressure | Time Frame: 30, 90, 180 and 365 days
  Change from baseline in systolic/diastolic blood pressure as indicated by average automated office blood pressure
Change in Systolic/Diastolic Blood Pressure - Ambulatory Blood Pressure Monitoring | Time Frame: 90, 180 and 365 days
  Change from baseline in systolic/diastolic blood pressure as indicated by ambulatory blood pressure monitoring
Effects on renal function assessed with glomerular filtration rate | Time Frame: 30, 90, 180 and 365 days
  Change from baseline in renal function as indicated by eGFR

CONTACTS AND LOCATIONS:
Locations (2):
- Georgia (2):
  - Israeli-Georgian Medical Research Clinic Helsicore, Tbilisi
  - Tbilisi Heart and Vascular Clinic, Tbilisi

IPD SHARING:
Plan to Share IPD: Undecided